CLINICAL TRIAL: NCT04859491
Title: Effects of Post-Exercise Recovery Drink Composition on Subsequent Performance in Masters Class Athletes
Brief Title: Effect of Carbohydrate-protein Co-ingestion on Short-term Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erica Goldstein (Other)
Responsible Party: Sponsor-Investigator, Erica Goldstein, Graduate Research Associate, University of Central Florida
Organization: University of Central Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MCAs and Short-Term Recovery
Record Dates: First submitted 2021-03-30; First posted 2021-04-26 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Dietary Supplementations
Keywords: glycogen; glucose; aerobic exercise; time to exhaustion; supplementation; protein; endurance; recovery
MeSH Terms: interventions — Carbohydrates

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of three groups: isocaloric carbohydrate (1.2 g/kg of body weight), carbohydrate-protein (0.8 g/kg body weight carbohydrate + 0.4 g/kg body weight protein), or placebo (flavored water). All three beverages will have a similar appearance and taste and participants will be blinded to the contents. All beverages will contain the same volume of fluid (1 liter).
Who Masked: Participant, Outcomes Assessor
Masking Description: The primary investigator will not be blinded to the treatment groups. However, both the research assistants responsible for administering the experimental protocol (aerobic interval and time to exhaustion testing) and the participants will be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbohydrate (Active Comparator): Carbohydrate in the amount of 1.2 g/kg of body weight (bw). Gatorade®, Chicago, IL, USA.
  Interventions: Dietary Supplement: Carbohydrate
- Carbohydrate-Protein (Active Comparator): Carbohydrate in the amount of 0.8 g/kg bw (Gatorade®, Chicago, IL, USA) plus protein in the amount of 0.4 g/kg bw (biPro Elite, Agropur Inc., Appleton, WI, USA).
  Interventions: Dietary Supplement: Carbohydrate-Protein
- Placebo (Placebo Comparator): Flavored water (G Zero, Gatorade®, Chicago, IL, USA).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Carbohydrate — Participants have a one in three chance of consuming a carbohydrate beverage between two bouts of high-intensity exercise.
  Other Names: CHO
  Arms: Carbohydrate
Dietary Supplement: Carbohydrate-Protein — Participants have a one in three chance of consuming a carbohydrate-protein beverage between two bouts of high-intensity exercise.
  Other Names: CHO-P
  Arms: Carbohydrate-Protein
Dietary Supplement: Placebo — Participants have a one in three chance of consuming a placebo beverage between two bouts of high-intensity exercise.
  Other Names: PLA
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the consumption of a carbohydrate, carbohydrate plus protein, or placebo sports drink during a 2-hour recovery period effectively moderates performance decrements during a subsequent bout of high-intensity exercise. This information will benefit any endurance-trained masters class athlete who may need to compete or train multiple times a day.

DETAILED DESCRIPTION:
To test the hypothesis, this study will utilize a randomized, double-blind, placebo-controlled between-subject design to examine the effects of carbohydrate (CHO) and carbohydrate-protein (CHO-P) supplementation on short-term recovery following aerobic interval exercise (INT) and time to exhaustion (TTE) testing in maters class athletes. After completing the informed consent and screening process (Visit #1), each participant will be assessed for their anthropometric measures as well as body composition and will complete a graded exercise test to volitional exhaustion on a cycle ergometer to determine VO2peak. Forty-eight to 72 hours after Visit #1, or VO2peak testing, participants will return to the lab for familiarization with the INT exercise protocol and TTE test (Visit #2). Within forty-eight to 72 hours after familiarization (Visit #2), participants will return to the lab for Visit #3 to complete INT exercise and TTE, a 2-hour passive recovery period including the consumption of one of three treatments (CHO, CHO-P, PLA), followed by repeated INT exercise and TTE, heart rate variability and sweat rate determination. Participants will also complete the Nutritional Recovery Practices, Knowledge, and Beliefs of Australian Triathletes survey during the 2-hour recovery period. Participants will be asked to complete the ASA24®, an automated self-administered 24-hour dietary assessment tool during the 5-9-day period between familiarization (Visit #2) and the experimental protocol (Visit #3).

ELIGIBILITY:
Inclusion Criteria:

* Men between the ages of 35 and 59 years
* Free of any physical limitations as determined by the Exercise Preparticipation Health Screening Questionnaire for Exercise Professionals (PHSQEP), and a Physical Activity Readiness Questionnaire for Everyone (PAR-Q+)
* Regularly engaged in endurance exercise (running, cycling, swimming) for a minimum of three years, a weekly training volume of 5-10 hours, and a maximal oxygen uptake of 45.00 ml·kg-1·min-1 or higher as determined by completion of VO2peak assessment (Visit #1).

Exclusion Criteria:

* Recent musculoskeletal injuries or surgeries
* Any chronic illness that requires continuous medical care
* Current incarceration, cognitive impairment or inability to provide consent
* Present or past use of performance-enhancing drugs

Ages: 35 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Time to Exhaustion (TTE) | Visit #3 (Day 7)
  Participants cycle for as long as possible at 90% of peak power output (watts)

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | Visit #3 (Day 7)
  R-R intervals recorded via a heart rate monitor and Elite HRV will be downloaded and analyzed using a laptop with commercially available HRV analysis software. Root mean square of the successive differences of R-R intervals (RMSSD) values will be recorded during the 90% TTE and then post-exercise every 5 min (end of TTE, 5min, 10min, 15min, 20min, 25min, 30min).
Sweat Rate (SR) | Visit #3 (Day 7)
  Sweat rate will be determined based on the difference between pre-and post-weight changes for each bout of exercise, the amount of fluid consumed during the recovery period, and total exercise time in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Stout, PhD, Study Chair — University of Central Florida; Erica Goldstein, MS, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCarthy DG, Spriet LL. Performance Effects of Carbohydrate Ingestion Between Bouts of Intense Aerobic Interval Exercise. Int J Sports Physiol Perform. 2020 Feb 1;15(2):262-267. doi: 10.1123/ijspp.2019-0239. Epub 2019 Jun 12. PMID 31188694
- [Result] Alghannam AF, Jedrzejewski D, Bilzon J, Thompson D, Tsintzas K, Betts JA. Influence of Post-Exercise Carbohydrate-Protein Ingestion on Muscle Glycogen Metabolism in Recovery and Subsequent Running Exercise. Int J Sport Nutr Exerc Metab. 2016 Dec;26(6):572-580. doi: 10.1123/ijsnem.2016-0021. Epub 2016 Aug 24. PMID 27097042
- [Result] Berardi JM, Price TB, Noreen EE, Lemon PW. Postexercise muscle glycogen recovery enhanced with a carbohydrate-protein supplement. Med Sci Sports Exerc. 2006 Jun;38(6):1106-13. doi: 10.1249/01.mss.0000222826.49358.f3. PMID 16775553

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT04859491/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT04859491/ICF_002.pdf